CLINICAL TRIAL: NCT00315796
Title: Nature Sights and Sounds to Reduce Pain in Cancer Patients Undergoing Bone Marrow Aspiration and Biopsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0387; NCCAM: AT00437
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2005-01

CONDITIONS: Cancer
Keywords: Mind-Body Intervention; Distraction; Biophilic; Cancer; pain; Bedscapes; procedures; bone marrow aspirate; bone marrow biopsy
MeSH Terms: conditions — Neoplasms; Pain

INTERVENTIONS:
Device: Biophilic Nature Scene and Sound

SUMMARY:
Pain is a common and difficult problem for patients with cancer. It has been reported that over 80% of cancer patients suffer from pain. Much of this pain is iatrogenic and related to procedures. Dr. Grossman recently demonstrated that most patients undergoing bone marrow biopsy have poor pain control during the procedure. Treatment of pain is almost entirely with analgesic medications, principally opioids. These medications have numerous undesirable effects such as sedation, confusion, hypotension and constipation that limit their efficacy and utility. Drs. Diette, Lechtzin, Rubin and colleagues recently demonstrated that use of nature sights and sounds (NSS), a simple, safe, and inexpensive intervention, decreases pain during fiberoptic bronchoscopy, a procedure commonly performed to diagnose cancer and to detect pulmonary complications of cancer therapy. Patients were randomly assigned to either standard care with intravenous narcotics and benzodiazepines or standard care coupled with view of a nature scene and use of nature sounds before, during, and after bronchoscopy. The group assigned to the NSS reported significantly better pain control than the control group. While these findings are novel and exciting, they raised several new questions that suggest logical extensions of this work. It is not known whether this intervention can be applied to patients in other settings, nor is it known whether comparison to standard care is an appropriate control group. Further, the mechanism of action of NSS needs to be determined. NSS may simply be a form of distraction therapy but it may have other properties. The theory of biophilia proposes there are specific elements in nature imagery that exert beneficial health effects. Because NSS appears to be a promising and safe intervention for the treatment of pain, these investigators plan to perform a controlled clinical trial in cancer patients undergoing invasive procedures. Patients will be randomly assigned to one of three arms, standard care, NSS, and a non-nature based distraction technique. We will study the efficacy of NSS for the management of procedure-related pain in oncology patients. The findings will provide necessary background information to develop more definitive studies of NSS that should be competitive for external funding. This exciting study will help develop a harmless, inexpensive method to treat pain in cancer patients, that may complement or replace analgesic medications.

DETAILED DESCRIPTION:
Study Design: This is a randomized, controlled trial assessing the impact of nature sights and sounds (NSS) on pain control in oncology outpatients undergoing bone marrow aspirate and biopsy (BMBx) in the Weinberg Cancer Center at Johns Hopkins. One hundred twenty patients will be assigned to one of three groups: 1) standard care, 2) NSS, 3) Music/Photo. The primary outcome will be pain scores during the procedures as measured by the Hopkins Pain Rating Instrument (HPRI). Patients in all groups will receive analgesic medications as dictated by the personnel performing the procedure and the physicians responsible for their clinical care. Patients in the NSS group will have Bedscapes nature scene murals placed at the bedside in a location that is visible throughout the procedure. They will also listen to a complementary audiotape during the procedure. The music/photo group will listen to city sounds during the procedure and view a poster of a city skyline.

Setting: The study will be conducted in the Weinberg Cancer Pavilion of the Kimmel Cancer Center at the Johns Hopkins Hospital.

Patient Selection: All patients 18 years and older with a diagnosis of cancer undergoing a BMBx in the Johns Hopkins Oncology Center will be screened for enrollment in the study.

Informed Consent: The study design and consent procedure will be explained to all prospective patients. If patients are interested in taking part in the study, written informed consent will be obtained. The study nurse will administer a mental status exam and assess eligibility. Consent and screening must occur within 5 days of the patient's procedure.

Randomization: Blocked randomization will be used with variable block sizes to ensure roughly equal numbers of patients in each study arm.

Study Interventions: All subjects will have pain managed by the physicians responsible for their clinical care as dictated by those physicians. Subjects assigned to NSS will have Bedscapes fabric panels depicting a scene of a mountain stream placed by the procedure table at a location where it will be visible throughout the procedure. An accompanying audiotape of complementary nature sounds will be played on portable tape players through headphones or speakers. They will be instructed to listen to the tape and look at the nature scene as frequently and for as long as they desire. The standard care group will have pain managed according to current oncology center protocols but will not be allowed to use the distraction interventions. The Music/Photo group will be played a tape of typical city sounds and will have a poster of a city skyline placed by the procedure table. The city skyline poster will be similar in size to the Bedscapes mural. The skyline image is a daytime photograph without water, trees or other nature elements. The subjects will be asked to listen to the music and view the picture during the procedure.

The HPRI will be used to measure pain. This is a plastic VAS with a sliding marker that moves within a grove. The side facing the patient appears like a traditional VAS. It has a 10cm line with the anchors "No Pain" and "Worst Pain Imaginable". The opposite side of the instrument is a 10 cm scale with markings every 0.5cm that enables the clinician to read and record numerical values (see figure in appendix). Scores will be recorded to the nearest 0.5cm. All patients will have a baseline assessment of pain immediately prior to the procedure. Subjects will be interviewed within one hour following the procedure and will be asked to quantify their pain during the procedure.Patients will also complete a questionnaire following the procedure in which they will score their level of pain control during the procedure on a 5-point Likert scale, which was used in the bronchoscopy study .

Data Collection: Following the procedure patients will complete a set of questionnaires. Questions will inquire about attitudes, beliefs and prior use of CAM. Patients in the NSS, and Music/Photo groups will be asked whether they found the study intervention to be helpful and if so what aspects of the intervention were beneficial. They will be asked to rate their satisfaction with several aspects of the procedure including comfort, the nursing care, the physician care, and the facility. Psychological distress will be measured with the Brief Symptom Index 18 , negative mood states and anxiety will be measured with the Profile of Mood States (POMS) . The BSI provides a global symptom severity score that will be used to control for subjects' underlying psychological distress, while POMS is well suited to measuring changes in mood related to the procedure. We will specifically focus on the Tension-Anxiety, Depression-Dejection, Anger-Hostility, and Confusion-Bewilderment subscales. Differences in response to pain will be measured with the Pain Catastrophizing Scale . Salivary cortisol will be measured before and after the procedure as a neuroendocrine marker of stress. Two baseline measurements of cortisol will be taken at least 15 minutes apart prior to the procedure. Immediately following the procedure three additional salivary cortisol samples will be collected approximately 15 minutes apart. The study nurse will record heart rate, blood pressure and respiratory rate before and every 15 minutes during the procedures. The high and low systolic blood pressure, heart rate, and respiratory rate will be extracted. The study nurse will record the percentage of time the patient used the study intervention during the procedure. Patients will also be asked what percentage of the time they used the intervention.

Outcomes: The primary outcomes is to determine if NSS is effective at reducing pain in cancer patients undergoing invasive procedures, we will compare mean pain scores during the procedure from the HPRI between the NSS group and the standard care group. We will also compare the difference between ratings of baseline pain and pain during the procedure in the two groups and the rating of pain control during the procedure between the groups. We will also determine if NSS reduces pain more than non-nature based distraction therapy we will compare pain ratings, and the difference in pain ratings from baseline to that during the procedure between the NSS and the music/photo group. Lastly we will determine if NSS reduces affective distress in cancer patients undergoing painful procedures we will compare mean scores from the POMS between the three groups. Secondary outcomes that pertain to all specific aims include vital signs during procedures and salivary cortisol levels. We will also assess overall satisfaction with care, ratings of physicians, ratings of nurses, and attitudes towards CAM interventions using Likert-type scales.

Sample Size: The primary outcome is difference in maximal pain level during procedures between the NSS group and the Music/Photo group. Power estimates are based on the magnitude of effect from the bronchoscopy study and the standard deviation of pain ratings in bone marrow biopsies studied by Dr. Grossman. In order to have 80% power to detect a 2-point difference in pain rating using the HPRI with an alpha error level of 0.05 we will need 29 patients in each group (total n=87). We plan to enroll 40 patients in each group (total n=120) to compensate for study withdrawal and missing data. We will continue to enroll patients until we have met these goals.

Data Entry and Management: The Biostatistics Core of the CAM center will provide recommendations on data entry and analysis. Because this is a small, single center trial of a relatively safe intervention there will not be a formal data safety monitoring committee. However, Dr. Lechtzin will oversee data integrity.

Adverse Events Monitoring: This is a minimal risk intervention and we expect very few adverse events. During our bronchoscopy study there was only one adverse event; a patient became incontinent on the procedure table due to the sound of running water. Adverse events to the experimental intervention will be assessed at the interview following the procedure by recording all voluntary complaints of subjects and through structured interviews. Attention will be directed to clinical adverse experiences associated with the procedure and the experimental intervention. In addition, all study participants will be provided a telephone number they can contact 24 hours/day, 7 days/week in case of questions, concerns, or adverse events. Adverse events will be documented on a standardized case report form. Summary reports of adverse events will be generated every three months. Dr. Lechtzin will review these. All serious adverse events including death, hospitalization, and premature withdrawal will be reported to the principal investigator within 24 hours of their occurrence. The principal investigator will report all serious adverse events to the Johns Hopkins IRB. Unexpected adverse events will be reported within 10 days.

Statistical Analysis: Analyses will be based on intention to treat. Analyses will be performed comparing patients who used NSS to the standard care group and the Music/Photo group. Descriptive analyses will be performed to assess subject characteristics (demographics, disease characteristics, education, prior CAM use and attitudes). Procedure characteristics will be compared including duration, complications, and medication usage. Continuous variables will be represented as mean plus or minus SE, medians and interquartile ranges. Bivariate analyses of outcomes will compare pain ratings, POMS subscales, and psychological distress between the groups. Chi squared test or Fisher's Exact test will be used to compare categorical variables such as age, gender, and race between groups. Unpaired t-tests or the Kruskal Wallis test will be used to compare continuous outcomes such as Pain Inventory scores. Pain scores will be analyzed as continuous variables and will also be categorized into mild (0-2), moderate (3-6) and severe (7-10). Multivariate analyses will be performed in order to adjust for possible confounding factors such as amount of narcotic analgesics given and amount of local anesthetic used. Ordinal logistic regression models to explain pain level by study intervention will be developed to adjust for factors such as age, gender, race, procedure type, education level, local anesthetic dose, narcotic dose, benzodiazepine dose, and BSI score. Additional factors will be included in the models if they are significant in bivariate analyses. Logistic regression models will be developed to determine factors associated with favorable response to NSS. Stepwise maximum-likelihood ratio estimation with a significance level of 0.2 for removal and 0.1 for inclusion will assist in model development. For all analyses significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Age>18
* Outpatient in the Weinberg Cancer Pavilion
* Capable of providing informed consent
* Undergoing bone marrow aspirate/biopsy
* Lack of any exclusion criteria

Exclusion Criteria:

* Visual impairment precluding use of nature scenes or city skyline photo
* Hearing impairment precluding use of compact discs or nature sounds
* Altered mental status (mental status score <25)
* Infection requiring contact isolation
* Language barrier that would limit ability to answer English language questionnaires
* Karnofsky performance score below 60
* Patients receiving conscious sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-08; Study Completion 2005-06

PRIMARY OUTCOMES:
Pain ratings: Hopkins Pain Rating Instrument

SECONDARY OUTCOMES:
Affective Distress: Profile of Moods States

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lechtzin, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lechtzin N, Busse AM, Smith MT, Grossman S, Nesbit S, Diette GB. A randomized trial of nature scenery and sounds versus urban scenery and sounds to reduce pain in adults undergoing bone marrow aspirate and biopsy. J Altern Complement Med. 2010 Sep;16(9):965-72. doi: 10.1089/acm.2009.0531. PMID 20799901